CLINICAL TRIAL: NCT06077903
Title: A Single Center, Single Arm Phase I Clinical Study of GT101 Injection in the Treatment of Metastatic/Recurrent Advanced Solid Tumors
Brief Title: GT101 Injection in the Treatment of Metastatic/Recurrent Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-FA-013
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GT101 treatment group (Experimental): Autologous tumor infiltrating lymphocyte injection
  Interventions: Biological: GT101

INTERVENTIONS:
Biological: GT101 — Autologous tumor infiltrating lymphocyte injection

SUMMARY:
This study is a single center, single arm phase I clinical trial. This study proposes to enroll 20 subjects, with a trial protocol including chemotherapy pretreatment, reinfusion of autologous tumor infiltrating lymphocyte injection, and interleukin-2 injection.

ELIGIBILITY:
Inclusion Criteria:

* 1. The Patients (or legally authorized representative) Patients (or legally authorized representative) must have the ability to understand the requirements of the study, have provided written informed consent as evidenced by signature on an informed consent form (ICF) approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC), must have the ability to understand the requirements of the study;
* 2.Must have a confirmed diagnosis of malignancy of their receptive histologies or cytologies: unresectable recurrent or metastatic solid tumor;
* 3.At least one resectable lesion (preferably superficial metastatic lymph nodes) that has not been treated with radiation and has not received other local therapies. The separated tissues mass Volume ≥1cm^3 (either of single lesion origin or multiple lesions combined) for the preparation of autologous tumor-infiltrating lymphocytes. Minimally invasive treatment where possible;

Exclusion Criteria:

* 1. Patients who have symptomatic and/or untreated CNS metastases (Except stable brain metastases, no medication required within 3 months, no hormone dependence);
* 2.Active infections requiring treatment with systemic anti-infectives (except for topical antibiotics); or those with unexplained fever > 38.5℃ occurring during the screening period, except for tumor fever;
* 3. Patients who have refractory or intractable epilepsy, active gastrointestinal bleeding or IL-2 contraindications;
* 4. Patients who have received allogeneic bone marrow transplantation or an organ allograft;
* 5.Patients who have a history of hypersensitivity to any component or excipient of study drugs: autologous tumor infiltrating lymphocytes, cyclophosphamide, fludarabine, IL-2, dimethyl sulfoxide (DMSO), human serum albumin (HSA), dextran-40 and antibiotics (beta lactam antibiotics, gentamicin);

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Incidience and severity of adversed events per CTCAE 5.0 | 3 years
  To characterize the safety profile of autologous TIL injection (GT101) in patients with relapsed/metastatic advanced solid tumor as measured by the incidience and severity of adversed events per CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No